CLINICAL TRIAL: NCT02946684
Title: Reducing the Impact of Ovarian Stimulation - The RIOT Project. Study RIOT-A: The Role of Aromatase Inhibitor in Reducing the Detrimental Effects of Ovarian Stimulation to Optimize Outcomes in Fresh Embryo Transfer Cycles
Brief Title: Effect of Addition of Aromatase Inhibitor to Ovarian Stimulation Therapy in IVF Treatment
Acronym: RIOT-A
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sven O. Skouby (Other)
Collaborators: Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Holbaek Sygehus (Other); Region Capital Denmark (Other); Copenhagen University Hospital, Denmark (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor-Investigator, Sven O. Skouby, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIOTA2015; 2015-005682-24 (EudraCT Number); H-15021850 (Other: Ethics Committee); HGH-2016-045_04513 (Other: Danish Data Protection Board)
Record Dates: First submitted 2016-07-11; First posted 2016-10-27 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Letrozole; Aromatase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactose Monohydrate (Placebo Comparator): 2 tablets of placebo are administered daily from stimulation start to day before hCG as adjunctive therapy to 150 IU of recFSH
  Interventions: Drug: Placebo
- Letrozole 5mg (Active Comparator): 2 tablets of 2,5mg Letrozole are administered daily from stimulation start to day before hCG as adjunctive therapy to 150 IU of recFSH
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Adjuvant therapy to recFSH during ovarian stimulation
  Other Names: Aromatase Inhibitor
  Arms: Letrozole 5mg
Drug: Placebo — Adjuvant therapy to recFSH during ovarian stimulation
  Other Names: Lactose Monohydrate
  Arms: Lactose Monohydrate

SUMMARY:
This project seeks to determine whether estradiol suppression achieved with adjuvant treatment with an aromatase inhibitor improves end-follicular and midluteal phase parameters during IVF. 128 patients will be randomized to either placebo or active treatment.

DETAILED DESCRIPTION:
The aim of the study is to investigate whether the detrimental effects of ovarian stimulation on outcomes in fresh embryo transfer cycles be ameliorated by co-treatment with aromatase inhibitors? The research questions are:

1. Can the impact of ovarian stimulation on late follicular phase sex steroid levels (and hence endometrial receptivity) be mitigated by co-treatment with aromatase inhibitors during ovarian stimulation?
2. Does co-treatment with aromatase inhibitors 'normalize' the endocrinology of the midluteal phase

ELIGIBILITY:
INCLUSION CRITERIA

* Indication for IVF/ICSI treatment
* Eligible for IVF/ICSI treatment according to local criteria
* Regular cycles 21-35 days (both included)
* Age < 40
* AMH 8- 32 (both included)
* Written consent

EXCLUSION CRITERIA

* Any contraindication for IVF/ICSI treatment according to local criteria
* Previous stimulation for IVF/ICSI with < 4 oocytes obtained
* PCOS
* Undergoing IVF/ICSI for the purpose of fertility preservation
* Allergy towards study drug

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Serum progesterone level | Assessed during stimulation treatment on day before hCG injection (throughout the study completion, up to 3 years)

SECONDARY OUTCOMES:
Serum estradiol, testosterone and androstenedione levels | Assessed on stimulation day 5, day of hCG administration (or the day before), day 7 and 10 after hCG administration. Assessed throughout study completion, up to 3 years.
P and 17-hydroxyprogesterone (17-HP) Area Under the Curve. | Assessed during stimulation treatment throughout the study completion, up to 3 years.
Follicular fluid concentration of estradiol, testosterone, inhibin B and AMH levels | Assessed during stimulation treatment (throughout the study completion, up to 3 years
Total IU of Follicle Stimulating Hormone used per cycle. | Assessed throughout study completion, up to 3 years
Number of follicles > 12 mm | Assessed in stimulated cycle on day of hCG administration or the day before (throughout the study completion), up to 3 years. Cycle length is between 21 and 35 days
Number of oocytes obtained oocytes obtained. | Assessed in stimulated cycle at time of oocyte pick up after follicle aspiration (throughout the study completion, up to 3 years).Cycle length is between 21 and 35 days
Proportion of oocytes resulting in top quality day 2, day 3 embryos or day 5/6 embryos according to validated morphological criteria. | Assessed at day 2-3 after oocyte pick up following stimulation (throughout study completion, up to 3 years)
Oocyte fertilization rate | Assessed during stimulation treatment (throughout the study completion, up to 3 years
Number and quality of embryos obtained, including rate of blastocyst formation. | Assessed during stimulation treatment (throughout the study completion, up to 3 years
Endometrial thickness in millimeters | Assessed throughout the study completion, up to 3 years
Implantation rate | Assessed during stimulation treatment (throughout the study completion, up to 3 years
Biochemical pregnancy rate | Assessed 2 weeks after embryo transfer following stimulation (throughout study completion, up to 3 years)
Clinical pregnancy rate | Pregnancy scan at gestational age week 7-8 (3-4 weeks after the positive hCG in serum). Assessed throughout study completion, up to 3 years.
Morphokinetic parameters of embryo quality as measured using a Time Lapse analysis in centers employing this technology. | Assessed from time of oocyte pick-up to embryo transfer following stimulation (throughout study completion, up to 3 years)
Reported side effects | From start of stimulation and administration of study medication to pregnancy scan week gestational age 7-8. Assessed throughout study completion, up to 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Sven O. Skouby, Professor, Principal Investigator — Unit of Reproductive Medicine, Herlev/Gentofte Hospital
Locations (4):
- Denmark (4):
  - Unit of Reproductive Medicine, Herlev Hospital, Herlev, Capital Region
  - Department of Fertility, Juliane Marie Centeret, Copenhagen, Capitol Region
  - Clinic of Fertility, Hvidovre Hospital, Hvidovre, Capitol Region
  - Clinic of Fertility, Holbæk Hospital, Holbæk, Region of Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bulow NS, Warzecha AK, Nielsen MV, Andersen CY, Holt MD, Petersen MR, Sopa N, Zedeler A, Englund AL, Pinborg A, Grondahl ML, Skouby SO, Macklon NS. Impact of letrozole co-treatment during ovarian stimulation on oocyte yield, embryo development, and live birth rate in women with normal ovarian reserve: secondary outcomes from the RIOT trial. Hum Reprod. 2023 Nov 2;38(11):2154-2165. doi: 10.1093/humrep/dead182. PMID 37699851
- [Derived] Bulow NS, Skouby SO, Warzecha AK, Udengaard H, Andersen CY, Holt MD, Grondahl ML, Nyboe Andersen A, Sopa N, Mikkelsen ALE, Pinborg A, Macklon NS. Impact of letrozole co-treatment during ovarian stimulation with gonadotrophins for IVF: a multicentre, randomized, double-blinded placebo-controlled trial. Hum Reprod. 2022 Jan 28;37(2):309-321. doi: 10.1093/humrep/deab249. PMID 34792133